CLINICAL TRIAL: NCT05789017
Title: Efficacy of Mycophenolate Mofetil Versus Leflunomide as Maintenance Treatment for IgG4-RD Patients With Internal Organ Involvement
Brief Title: Treatment Strategies for IgG4-RD Patients With Internal Organ Involvement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Wen Zhang, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Management for IgG4-RD
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Autoimmune Diseases
Keywords: Immunoglobulin G4-Related Disease; treatment strategies; relapse; leflunomide; mycophenolate mofetil
MeSH Terms: conditions — Autoimmune Diseases; Immunoglobulin G4-Related Disease; Recurrence | interventions — Prednisone; Mycophenolic Acid; Leflunomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): Patients are treated with glucocorticoids and mycophenolate mofetil in remission induction period (6 months), during which glucocorticoids are tapered regularly and discontinued in 6 months. Afterwards, patients are treated with low dose mycophenolate (1-1.5g/day) during remission maintenance period for 12 months.
  Interventions: Drug: Prednisone and Mycophenolate Mofetil; Drug: Mycophenolate Mofetil
- Group II (Experimental): Patients are treated with glucocorticoids and mycophenolate mofetil in remission induction period (6 months), during which glucocorticoids are tapered regularly and discontinued in 6 months. Afterwards, patients are treated with leflunomide (20 mg/day) during remission maintenance period for 12 months.
  Interventions: Drug: Prednisone and Mycophenolate Mofetil; Drug: Leflunomide

INTERVENTIONS:
Drug: Prednisone and Mycophenolate Mofetil — Patients are treated with glucocorticoids and mycophenolate mofetil in remission induction period (6 months), during which glucocorticoids are tapered regularly and discontinued in 6 months.
Drug: Mycophenolate Mofetil — Patients are treated with low dose mycophenolate (1-1.5g/day) during remission maintenance period for 12 months.
  Arms: Group I
Drug: Leflunomide — Patients are treated with leflunomide (20 mg/day) during remission maintenance period for 12 months.
  Arms: Group II

SUMMARY:
This study has been designed as a 18-month, open-label randomized controlled clinical trial. The study aims to compare the efficacy and safety of two treatment strategies in active IgG4-RD patients with internal organ involvement during maintenance remission period: low dose mycophenolate mofetil group and leflunomide group.

DETAILED DESCRIPTION:
60 active IgG4-RD patients with internal organ involvement are enrolled in this study and accept the combination treatment of glucocorticoids and mycophenolate mofetil in remission induction period (6 months), during which glucocorticoids are tapered regularly and discontinued in 6 months. During remission maintenance period, pateints are randomly divided into two groups at a 1:1 ratio: patients in group I are treated with low dose mycophenolate mofetil (1-1.5g/day) and patients in group Ⅱ accept the treatment of leflunomide (20 mg/day). Patients in two groups will be followed up for another 12 months, and clinical evaluations, laboratory tests, image examinations and IgG4-RD responder index (RI) will be recorded during follow up. The primary endpoint is the difference of relapse rate between two groups at 18 months. The secondary endpoints are relapse time, response rate and side effects.

ELIGIBILITY:
Inclusion Criteria:

* 1. Fulfillment of the 2019 American College of Rheumatology/European League against Rheumatology (ACR/EULAR) IgG4-related disease classification criteria; 2. Newly-onset or relapsed patients who requires initiation or continuation of glucocorticoids treatment.

Exclusion Criteria:

* 1. Patients who were diagnosed as other autoimmune diseases; 2. Patients who were diagnosed as malignant diseases; 3. Pregnant and lactating women； 4. Active infection: HIV, HCV, HBV, TB； 5. Severe irreversible damage of organ function; 6. Receipt of any biologic therapy or immunosuppressive agent other than GCs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The difference of relapse rate of IgG4-RD between two groups in 18 months. | 18 months
  The definition of relapse: elevation of IgG4-RD Responder Index ≥ 2 points; new organ involvement or recurrence, with or without elevation of serum IgG4 levels.

SECONDARY OUTCOMES:
The difference of the time at baseline to first relapse between two groups. | 18 months
Response rate to the treatment of the two groups. | 18 months
  Complete response rate; Partial response rate; No response
Side effects | 18 months
  Any side effects caused by treatments for IgG4-RD.

CONTACTS AND LOCATIONS:
Overall Officials: Wen Zhang, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China